CLINICAL TRIAL: NCT02431858
Title: Catheter Over Needle Technique Causes Less Leakage and Secondary Failure Than Catheter Through Needle Technique for Continuous Femoral Nerve Block
Brief Title: Catheter Over Needle vs Catheter Through Needle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Charles Gairdner Hospital (Other)
Responsible Party: Principal Investigator, Richard Edwards, Principle Investigator, Sir Charles Gairdner Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-011
Record Dates: First submitted 2015-04-22; First posted 2015-05-01 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Nerve Block; Catheterization
Keywords: Nerve block; Catheter; Catheter over needle; Femoral Nerve; Anaesthesia; [E04.525.210.550]; [E02.148]

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter Over Needle (Experimental): The femoral nerve catheter used will be the "E-Catheter" (Pajunk) device which is a novel catheter over needle system.
  Interventions: Device: E-Catheter (Pajunk)
- Catheter through needle (Active Comparator): The femoral nerve catheter used will be the "Sonolong" catheter (Pajunk) which is a traditional catheter through needle system.
  Interventions: Device: Sonolong Catheter (Pajunk)

INTERVENTIONS:
Device: E-Catheter (Pajunk)
  Other Names: Australian Therapeutic Goods Registry (ATGR) no: 133630
  Arms: Catheter Over Needle
Device: Sonolong Catheter (Pajunk)
  Other Names: Australian Therapeutic Goods Registry (ATGR) no: 133630
  Arms: Catheter through needle

SUMMARY:
To randomize 108 patients undergoing knee replacement surgery to catheter through needle or catheter over needle femoral nerve blocks, then monitor the catheters for leakage to see if there is a difference.

DETAILED DESCRIPTION:
Background: Total Knee Replacement Surgery is a commonly performed procedure that causes significant post-operative pain. Continuous femoral nerve blocks are widely used for analgesia as part of a multimodal analgesic regimen for this surgery. They provide sustained analgesia which allows early physiotherapy for rehabilitation. Currently the most common technique for inserting catheters for continuous femoral nerve blocks is to feed a catheter though a needle (CTN) which has been placed close by the nerve. There is a significant rate of leak and dislodgement of these catheters which can lead secondary failure where the catheter is no longer providing analgesia by blocking the nerve (primary failure occurs when the nerve block catheter fails to provide any analgesia from the start). The system to be investigated has a catheter over the needle (CON) which is left in place after the needle is withdrawn. The proposed benefit of this is that there will be a reduction in leak rates and dislodgement. This is because using a CON technique means that the biggest hole will be the diameter of the catheter, rather than CTN where the biggest hole will be the diameter of the needle therefore allowing leak around the outside of the catheter.

Objectives: To ascertain whether or not the catheter over needle technique is superior to catheter through needle technique in terms of a leak rate.

Trial plan: To recruit 108 patients who are having total knee replacement surgery into the study and randomise them into having either CON or CTN continuous femoral nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Sir Charles Gairdner Hospital for elective, unilateral, primary total knee replacement.
* Body mass index 18-40 kg/m2
* American Society of Anaesthetists (ASA) grade I-III

Exclusion Criteria:

* Allergy to local anaesthetic
* Inability to cooperate
* Inability to read, speak and understand English
* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Catheter leakage | 2 days post insertion
  Any leakage around the catheter insertion site as assessed by visual inspection.

SECONDARY OUTCOMES:
Overall rate of secondary failure as assessed by the acute pain service on days 1 and 2 post op. | 2 days
  Secondary failure is when a nerve catheter that was previously working has ceased to provide analgesia.
Ease of insertion assessed by the inserting anaesthetist on a 5 point Likert scale. | intraoperative
  Assess the anaesthetist's opinion on the ease of insertion of the different catheters
Needle visibility assessed by the inserting anaesthetist on a 5 point Likert scale. | intraoperative
  Assessing the needle visibility in the two different catheter systems.

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Edwards, MBBS, Principal Investigator — Sir Charles Gairdner Hospital
Locations (1):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia